CLINICAL TRIAL: NCT07034924
Title: Temporary Aortic Compression With the Abdominal Tourniquet for Refractory Postpartum Hemorrhage
Acronym: ACT-PPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LLC UkrMedGroup (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/EC/15051
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, interventional treatment study designed to assess the effectiveness and safety of the AAJT-S device in the management of severe postpartum hemorrhage. All eligible participants will receive the same intervention without randomization or control group. Data will be collected in real time across multiple centers, and the study does not include blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Participant Group/Arm (Experimental): Participants in this arm will receive standard postpartum hemorrhage (PPH) management followed by application of the Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) device if bleeding remains uncontrolled after uterotonics and uterine balloon tamponade. The device will be applied to the upper abdomen and inflated to 250 mmHg to achieve temporary aortic occlusion for up to 60 minutes. The intervention is intended to temporize bleeding while definitive surgical treatment and blood transfusion are arranged.
  Interventions: Device: Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S)

INTERVENTIONS:
Device: Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) — The AAJT-S is a non-invasive, externally applied medical device designed to achieve temporary occlusion of the abdominal aorta and inferior vena cava by inflating a pneumatic bladder to 250 mmHg. In this study, the device will be used as a temporizing measure for patients with severe postpartum hemorrhage unresponsive to standard uterotonics and balloon tamponade. The device will be applied horizontally over the upper abdomen and inflated using a built-in pressure gauge. The intended effect is to reduce pelvic blood flow and allow time for mobilization of surgical resources and blood transfusion. Maximum application time will not exceed 60 minutes, in accordance with established safety guidelines.

SUMMARY:
This multicenter study aims to evaluate effectiveness and safety of using the AAJT-S device as a temporary intervention for severe, atony-related PPH that is refractory to standard therapies

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm treatment study aimed at evaluating the feasibility, safety, and clinical effectiveness of the Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) as a temporary intervention for managing severe postpartum hemorrhage (PPH) caused by uterine atony unresponsive to standard first-line treatments. The study will be conducted across several sites in Ukraine, in regions affected by armed conflict, where access to surgical care and blood products may be delayed.

Eligible participants are postpartum women aged 18 or older who experience primary PPH with estimated blood loss greater than 1000 mL and who do not respond to uterotonics or balloon tamponade. Patients with hemorrhage due to trauma, coagulopathy, or retained placental tissue will be excluded.

When standard interventions fail and eligibility is confirmed, the AAJT-S device will be applied to the upper abdomen and inflated to 250 mmHg to temporarily occlude the abdominal aorta and inferior vena cava. This intervention aims to reduce pelvic blood flow and control bleeding, buying critical time to assemble the surgical team, initiate blood transfusion, and establish anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of postpartum hemorrhage (PPH) refractory to uterotonics and intrauterine balloon tamponade
* Estimated blood loss greater than 1300 mL
* Oral informed consent provided prior to device application

Exclusion Criteria:

* Patients with postpartum bleeding as a result of trauma, retained placenta or coagulopathy were excluded

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy: The proportion of cases achieving rapid hemorrhage control after AAJT-S application. | Within 5 minutes of AAJT-S device application
  Visible cessation of external vaginal bleeding (no ongoing blood flow from the cervix or vaginal canal observed by the clinical team) within 5 minutes of device inflation. The attending obstetrician will visually assess bleeding immediately after inflation and every 30 seconds until 5 minutes. "Control" will be recorded at the first time point when no active bleeding is observed (slight spotting is not considered ongoing hemorrhage). If bleeding persists beyond 5 minutes, the case is classified as "failure of primary endpoint," even if subsequent control is achieved.
Safety: Incidence (i.e., Rate or Number of Participants), Severity and Seriousness of Device-related Adverse Events from placement until 6-week postpartum follow-up | From device application until 6-week postpartum follow-up
  Any untoward medical occurrence temporally associated with the AAJT-S device, regardless of causality

SECONDARY OUTCOMES:
Visually estimated blood loss (EBL) | From delivery until AAJT-S placement
  Visually estimated blood loss (EBL) from delivery until AAJT-S placement (mL).

CONTACTS AND LOCATIONS:
Overall Officials: Yevheniia Poliakova, Ph.D, Principal Investigator — LLC UkrMedGroup
Locations (1):
- Olexandrivska Hospital, Zaporizhzhia, Ukraine

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and the sensitive nature of the clinical context, including emergency obstetric care in a war-affected setting. Additional ethical and regulatory considerations related to patient privacy and consent limit the possibility of external data sharing.

REFERENCES:
- [Background] Khan M, Jeyanathan J, Smith JE. Novel use for the abdominal tourniquet in the management of postpartum haemorrhage. J R Army Med Corps. 2018 Nov;164(6):463. doi: 10.1136/jramc-2018-000953. Epub 2018 Apr 6. No abstract available. PMID 29626141
- [Background] Nieto-Calvache AJ, Palacios Jaraquemada JM, Basanta N, Aryananda RA, Sinisterra-Diaz SE, Rodriguez F, Hidalgo Cardona A, Messa Bryon A. Internal manual compression of the aorta-an effective way to temporarily control pelvic bleeding in obstetrical hemorrhage. Am J Obstet Gynecol. 2022 Jul;227(1):96-97. doi: 10.1016/j.ajog.2022.02.040. Epub 2022 Mar 4. PMID 35248574
- [Background] Riley DP, Burgess RW. External abdominal aortic compression: a study of a resuscitation manoeuvre for postpartum haemorrhage. Anaesth Intensive Care. 1994 Oct;22(5):571-5. doi: 10.1177/0310057X9402200512. PMID 7818062
- [Background] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Aryananda RA, Basanta N, Cininta N, Rivera-Torres LF, Bautista E, Hussein AM. External aortic compression: buying time to save lives in obstetric hemorrhage. Am J Obstet Gynecol. 2025 Feb;232(2):239-241. doi: 10.1016/j.ajog.2024.09.017. Epub 2024 Sep 18. No abstract available. PMID 39304012
- [Background] Kheirabadi BS, Dubick MA. Safe duration of Abdominal Aortic and Junctional Tourniquet application. J Trauma Acute Care Surg. 2019 Sep;87(3):740-741. doi: 10.1097/TA.0000000000002231. No abstract available. PMID 30768561
- [Background] Soltan MH, Faragallah MF, Mosabah MH, Al-Adawy AR. External aortic compression device: the first aid for postpartum hemorrhage control. J Obstet Gynaecol Res. 2009 Jun;35(3):453-8. doi: 10.1111/j.1447-0756.2008.00975.x. PMID 19527382
- [Background] Soltan MH, Sadek RR. Experience managing postpartum hemorrhage at Minia University Maternity Hospital, Egypt: no mortality using external aortic compression. J Obstet Gynaecol Res. 2011 Nov;37(11):1557-63. doi: 10.1111/j.1447-0756.2011.01574.x. Epub 2011 Jun 16. PMID 21676082
- See also: Information about The Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) — https://www.narescue.com/abdominal-aortic-and-junctional-tourniquet-stablized-aajt-s.html